CLINICAL TRIAL: NCT01376570
Title: A Randomized Trial of an Abstinence-reinforcing Contingency Management Intervention to Suppress HIV Viral Load
Brief Title: Project FIRST - Financial Incentives to Reduce Substance Use and Improve Treatment
Acronym: Project FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Chinazo Cunningham, Associate Professor of Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-553; R01DA032110 (NIH)
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: HIV; Opiate Dependence
Keywords: HIV; Opiate dependence; Opiate replacement therapy; Cocaine-related disorders; Risk Reduction Behavior; Medication Adherence; Motivation
MeSH Terms: conditions — Opioid-Related Disorders; Cocaine-Related Disorders; Risk Reduction Behavior; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contingency Management arm (Experimental): The Contingency Management arm will receive the abstinence-reinforcing contingency management intervention.
  Interventions: Behavioral: Abstinence-reinforcing contingency management intervention
- Control arm (Active Comparator): The Control arm will receive the performance feedback intervention.
  Interventions: Behavioral: Performance Feedback intervention

INTERVENTIONS:
Behavioral: Abstinence-reinforcing contingency management intervention — The contingency management intervention consists of participants receiving vouchers exchangeable for goods and services contingent on achieving abstinence. When participants are abstinent (urine is free of cocaine, oxycodone and opiates), they will receive a voucher. If participants are not abstinent (cocaine or oxycodone or opiates are in the urine), they will not receive a voucher. The value of vouchers increases with continued evidence of abstinence. When participants have urines with opiates or cocaine, the value of the voucher is reset. The vouchers are part of the intervention, they are not participant compensation.
  Arms: Contingency Management arm
Behavioral: Performance Feedback intervention — Participants will receive performance feedback about their drug use. The research team will provide informational slips of paper indicating results of urine tests and will congratulate participants when urines are drug-free or encourage participants to stop using cocaine and/or opiates when urines are not drug-free.
  Arms: Control arm

SUMMARY:
This study will test whether contingency management (monetary vouchers contingent on abstinence from drugs) that reinforces one behavior (achieving abstinence from drugs) leads to improved outcomes in other related behaviors (achieving HIV viral load suppression). In a randomized controlled trial, the investigators propose to test whether an abstinence-reinforcing contingency management intervention improves viral load suppression in HIV-infected drug users.

DETAILED DESCRIPTION:
Using a randomized controlled study design, the investigators will test the efficacy of an abstinence-reinforcing contingency management intervention compared with a control condition (Performance Feedback) on HIV viral load suppression. The investigators will enroll 202 opioid-dependent HIV-infected individuals who are receiving opioid agonist treatment with buprenorphine or methadone, who continue to use opiates, oxycodone or cocaine (drugs that are consistently associated with poor HIV treatment outcomes), and who are prescribed antiretroviral medication, but with suboptimal viral load suppression. The contingency management group will have the potential to receive compensation in vouchers over the 16-week intervention based on drug-free urine. Participants will be followed for 28 weeks, with research visits occurring twice weekly during the Baseline Period (weeks 1-4) and Intervention Period (weeks 5-20), then every two weeks during the Post-Intervention Period (weeks 21-28). Data sources will include blood tests (viral load and CD4 count), urine toxicology tests, questionnaires, pill counts, and medical records. The primary outcome will be change in HIV viral load, and secondary outcomes will include CD4 count, antiretroviral adherence, and abstinence.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* English or Spanish fluency
* HIV-infected
* Currently taking highly active antiretroviral therapy
* a) opioid use disorder and receiving opioid agonist treatment with methadone or buprenorphine, or b) cocaine use disorder
* urine toxicology positive for cocaine, oxycodone, or opioids during the run-in period
* detectable viral load while prescribed highly active antiretroviral therapy in the prior 6 months
* self-reported adherence to HAART <100%

Exclusion Criteria:

* inability to give informed consent
* inability to follow the research protocol (e.g., visits twice weekly)
* frequent hospitalizations (>2) in the prior 6 months
* currently with a chronic pain condition in which the participant has been prescribed opioid analgesics for longer than the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2012-06; Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
HIV viral load | Viral load will be measured every 4 weeks over the 28-week follow-up period.
  Every 4 weeks participants will undergo phlebotomy to measure HIV viral load. Viral load will be analyzed as a continuous measure (log10 copies/ml). In secondary analyses, viral load will be analyzed dichotomously, as undetectable (<45 copies/ml) or not.

SECONDARY OUTCOMES:
CD4 count | CD4 count will be measured at weeks 0, 4, 20, and 28.
  At weeks 0, 4, 20, and 28, participants will undergo phlebotomy and CD4 count will be measured. CD4 count will be analyzed as a continuous measure and an increase of 50 cells/mm3 will be considered a clinically significant improvement.
Abstinence from opiates, oxycodone, and cocaine | Abstinence will be measured twice weekly during weeks 0-20, then every two weeks during weeks 21-28.
  Participants will provide urine samples twice weekly during weeks 0-20, and every two weeks during weeks 21-28. Abstinence will be defined as having drug-free urine (no cocaine, oxycodone and opiates). Abstinence will be examined two different ways-as the proportion of drug-free urines and the number of consecutive drug-free urines. Although urine toxicology tests will be our primary data source for measuring abstinence, we will also measure addiction severity using the Addiction Severity Index.
Antiretroviral adherence | Antiretroviral adherence will be measured every 4 weeks during the 28-week follow-up period
  Antiretroviral adherence will be measured using pill counts. Adherence will be analyzed as a continuous measure, defined as the proportion of pills taken (# pills taken / # pills prescribed). Mean adherence over each 4-week period will be examined. In addition, we will also analyze adherence as a dichotomous measure (e.g., perfect [100%] adherence or not during each 4-week period).

CONTACTS AND LOCATIONS:
Overall Officials: Chinazo Cunningham, MD,MS, Principal Investigator — Albert Einstein College of Medicine
Locations (3):
- United States (3):
  - Montefiore's Community Clinics (Montefiore Medical Group), The Bronx, New York
  - Albert Einstein College of Medicine Division of Substance Abuse clinics, The Bronx, New York
  - Montefiore Infectious Disease Clinic, The Bronx, New York

REFERENCES:
- See also: Abstinence-reinforcing contingency management improves HIV viral load suppression among HIV-infected people who use drugs: A randomized controlled trial — https://doi.org/10.1016/j.drugalcdep.2020.108230